CLINICAL TRIAL: NCT05833763
Title: An Open-label, Single-arm, Phase 2 Trial of GlOfitamab anD pIrtobrutinib (LOXo-305) in Patients With Mantle Cell Lymphoma and Prior Exposure to a BTK Inhibitor
Brief Title: A Phase 2 Trial of GlOfitamab anD pIrtobrutinib in Mantle Cell Lymphoma Patients With Prior BTK Inhibitor Exposure.
Acronym: GOlDiLOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Leukaemia and Lymphoma Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHL37
Record Dates: First submitted 2023-03-26; First posted 2023-04-27 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Mantle Cell Lymphoma; Mantle Cell Lymphoma Refractory
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — glofitamab; pirtobrutinib; obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Treatment (Experimental): This study design involves 3 phases:
  1. Treatment Ramp-Up
     1. Pre-Phase (7 days): Obinutuzumab (1000mg) will be administered intravenously (IV) on D-7 and a second dose administered between Day 6 and Day 1.
     2. Cycle 1: An initial dose level of Glofitamab will evaluate step-up dosing. If excessive dose-limiting toxicity is observed, including cytokine release syndrome (CRS), a lower initial dose of 1.25mg of glofitamab will be evaluated at "dose level -1".
     i. Dose level 1 (14 days):
     * 2.5mg Glofitamab by IV on Day 1
     * 10mg Glofitamab by IV on Day 8 ii. Dose level -1 (21 days):
     * 1.25mg Glofitamab by IV on Day 2
     * 2.5mg Glofitamab by IV on Day 8
     * 10mg Glofitamab by IV on Day 15 c. Cycle 2 (21 days): 30mg Glofitamab by IV on Day 1
  2. Fixed course combination phase: Cycles 3-12 (21 days per cycle): 30mg of Glofitamab by IV on day 1
  3. Maintenance phase: Cycles 13+ (21 days per cycle): Glofitamab discontinued. 200mg oral daily
  Interventions: Drug: Glofitamab; Drug: Pirtobrutinib; Drug: Obinutuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab is provided as liquid concentrate for IV infusion. Each vial contains 10mg of glofitamab.
Drug: Pirtobrutinib — Pirtobrutinib is supplied as immediate release film-coated tablets containing 50 mg, or 100 mg of active compound. Tablets are supplied in labelled, HDPE bottles and sealed with child-resistant closures.
Drug: Obinutuzumab — Obinutuzumab is provided as a single dose 1000 mg liquid concentrate for infusion containing of 25 mg/mL obinutuzumab.
Drug: Tocilizumab — Tocilizumab is provided as a liquid concentrate for IV infusion. Each vial contains 200mg/10mL concentrate solution

SUMMARY:
The goal of this clinical trial is to evaluate the safety and response of combining Pirtobrutinib and Glofitimab in patients with relapsed MCL. The main question it aims to answer are:

* Will additive and synergistic effects be observed when using a combination of glofitamab and pirtobrutinib?
* Will this combination be safe and lead to high complete- and remission rates with no residual disease?

Pirtobrutinib will be given to all participants as an oral tablet for the duration of the entire study. Participants will receive other treatment in 3 phases:

1. Treatment Ramp-Up

   1. Treatment with Obinutuzumab by Intravenous (IV)
   2. An initial dose level of Glofitamab will evaluate step-up dosing. If excessive adverse events are observed, a lower initial dose will be used.
2. Fixed course combination phase: Treatment with Glofitamab by IV
3. Maintenance phase: Glofitamab is discontinued. 200mg oral daily

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the safety and response of combination Pirtobrutinib and Glofitimab in patients with relapsed/refractory MCL. The main question it aims to answer are:

* Will additive and synergistic effects be observed when using a combination of glofitamab and pirtobrutinib?
* Will this combination be safe and lead to high complete- and MRD-negative remission rates?

Participants will receive treatment based on 21 day cycles. This study design involves 3 phases:

1. Treatment Ramp-Up

   1. Pre-Phase (7 days): Obinutuzumab (1000mg) will be administered intravenously (IV) on D-7 and a second dose administered between Day 6 and Day 1.
   2. Cycle 1: An initial dose level of Glofitamab will evaluate step-up dosing. If excessive dose-limiting toxicity is observed, including cytokine release syndrome (CRS), a lower initial dose of 1.25mg of glofitamab will be evaluated at "dose level -1".

   i. Dose level 1 (14 days):
   * 2.5mg Glofitamab by IV on Day 1
   * 10mg Glofitamab by IV on Day 8 ii. Dose level -1 (21 days):
   * 1.25mg Glofitamab by IV on Day 2
   * 2.5mg Glofitamab by IV on Day 8
   * 10mg Glofitamab by IV on Day 15 c. Cycle 2 (21 days): 30mg Glofitamab by IV on Day 1
2. Fixed course combination phase: Cycles 3-12 (21 days per cycle): 30mg of Glofitamab by IV on day 1
3. Maintenance phase: Cycles 13+ (21 days per cycle): Glofitamab discontinued. 200mg oral daily

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 years old or above
2. A confirmed diagnosis of MCL according to World Health Organization (2016) criteria
3. At least one site of measurable disease not previously irradiated (defined as at least one bi-dimensionally measurable nodal lesion of greater than or equal to 1.5cm in longest dimension)
4. Life expectancy (in the opinion of the investigator) of greater than or equal to 18 weeks
5. Prior therapy with a BTK inhibitor alone or in combination and:

   1. Progression or relapse post BTK inhibitor or
   2. Failed to achieve PR following 12 weeks of BTK inhibitor therapy
6. Prior TRAEs must have recovered to Grade 1 or less with the exception of alopecia, peripheral neuropathy and lymphopenia.
7. ECOG 0-2
8. Adequate washout of prior therapies:

   1. Broad field radiation (greater than or equal to 30% of the bone marrow or whole brain radiotherapy) must be completed 14 days prior to study treatment
   2. Palliative limited field radiation must be completed 7 days prior to study treatment.
   3. Targeted agents, investigational agents, therapeutic monoclonal antibodies/antibody drug conjugates or cytotoxic chemotherapy must be completed 5 half-lives or 2 weeks (whichever is shorter) prior to study treatment (except for BTK inhibitors which may be continued until 1 day prior to planned first therapy with pirtobrutinib)
   4. Steroids (prednisolone less than or equal to 100mg daily or equivalent for up to 14 days are permitted during screening for control of lymphoma related symptoms
9. Ability to take oral medications
10. Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
11. Willingness of men and women of reproductive potential to observe conventional and highly effective and acceptable birth control methods for the duration of treatment and for six months following the last dose of study treatment
12. Women of childbearing potential must have a negative serum pregnancy test within seven days of enrolment
13. Adequate coagulation, defined as aPTT and PT not greater than 1.5xULN, unless laboratory abnormality is explained by concomitant anticoagulant medication, a lupus anticoagulant, or a factor deficiency not associated with an increased bleeding risk, as determined by the investigator.
14. Adequate liver function:

    * ALT and AST less than or equal to 3X ULN, or less than or equal to 5X ULN if documented liver involvement
    * Total bilirubin less than or equal to 1.5X ULN or less than or equal to 5X ULN if documented liver involvement and/or Gilbert's Disease
15. Adequate renal function

    - Creatinine clearance greater than or equal to 30mls/minute according to Cockroft-Gault formula
16. Adequate haematological parameters

    * Haemoglobin greater than or equal to 80g/L (transfusion support permitted)
    * Absolute neutrophil count greater than or equal to 1.0x10^9/L (May be G-CSF supported)
    * Platelets greater than or equal to 75 X 10^9/L. OR platelets greater than or equal to 50 X 10^9/L if documented marrow involvement or splenomegaly (must be platelet transfusion independent for 7 days prior to first dose of obinutuzumab
17. Sufficient archival tissue is available for central review or after discussion with the CPI

Exclusion Criteria:

1. Inability to comply with protocol mandated hospitalisations
2. For patients enrolling on the safety cohort, a history of allogeneic transplantation within 12 months of enrolment or ongoing chronic GVHD or immunosuppressive therapy.
3. Autologous SCT or CAR-T therapy within 6 weeks of enrolment
4. Active central nervous system involvement with MCL
5. Prior treatment with pirtobrutinib or demonstrated refractoriness to a CD20xCD3 bispecific antibody.
6. Have a known severe hypersensitivity to any of the excipients of pirtobrutinib, glofitamab, tocilizumab or obinutuzumab.
7. History of stroke or intracranial haemorrhage within six months of enrolment.
8. Live vaccination within 28 days of enrolment.
9. Major surgery or significant traumatic injury within 28 days of study treatment or the anticipation of major surgery during study treatment (surgical procedures for the diagnosis of lymphoma such as lymph node resection/ laparoscopy are allowed provided patient is considered fit for treatment as judged by investigator)
10. Significant cardiovascular disease defined as:

    1. Unstable angina or acute coronary syndrome within 2 months of registration
    2. History of myocardial infarction within 3 months prior to registration
    3. Documented LVEF by any method of = 40% during screening
    4. Grade 3 or higher NYHA functional classification system of heart failure
    5. Uncontrolled or symptomatic arrhythmias
11. Prolongation of the QT interval corrected for heart rate (QTcF) greater than 470 msec on at least 2/3 consecutive electrocardiograms (ECGs), and mean QTcF greater than 470 msec on all 3 ECGs, during Screening. QTcF is calculated using Fridericia's Formula (QTcF): QTcF euqal to QT/(RR0.33) Correction of suspected drug-induced QTcF prolongation can be attempted at the investigator's discretion and only if clinically safe to do so with either discontinuation of the offending drug or switching to another drug not known to be associated with QTcF prolongation. Correction for underlying bundle branch block (BBB) allowed. Patients with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias
12. Known human immunodeficiency virus (HIV) infection
13. Known active HBV or HCV infection based on criteria below:

    1. HBV: Patients with positive HbsAg are excluded. Patients with positive hepatitis B core antibody antiHBc and negative HbsAg require negative hepatitis B PCR before enrolment and must be treated with antiviral therapy. Patients who are hepatitis B PCR positive will be excluded.
    2. HCV: If positive hepatitis C antibody, patient will need to have a negative hepatitis C RNA before enrolment. Patients who are hepatitis C RNA positive will be excluded.
14. Known active CMV infection. Unknown or negative status are eligible.
15. Pregnancy, lactation or plan to breastfeed during the study or within 6 months of the last dose of study treatment.
16. Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of pirtobrutinib.
17. Evidence of other clinically significant uncontrolled condition(s) including but not limited to, uncontrolled systemic bacterial, viral, fungal or parasitic infection, or other clinically significant active disease process which in the opinion of the investigator and medical monitor may pose a risk for patient participation.
18. Active uncontrolled auto-immune cytopenia (e.g., AIHA, ITP) for which new therapy was introduced or existing therapy was escalated within the 4 weeks prior to study enrolment to maintain adequate blood counts, unless auto-immune cytopenias are secondary to MCL
19. Active second malignancy unless in remission and with life expectancy greater than 2 years.
20. Current treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers and/or strong P-gp inhibitors.
21. Patients requiring therapeutic anticoagulation with warfarin or another vitamin K antagonist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2032-04 (Estimated); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of combination Pirtobrutinib and Glofitmab in patients with relapsed/refractory MCL and prior BTK inhibitor exposure. | Following six cycles (or approximately 18 weeks following first treatment). Cycle 1 is 14 days in duration and cycles 2 to 6 are 21 days in duration.
  Determined by the complete response (CR) rate according to Lugano criteria

SECONDARY OUTCOMES:
Complete response rate using the Lugano Criteria for response assessment at end of 12 cycles of Glofitamab | When all patients have completed 12 cycles of Glofitamab. Cycle 1 is 14 days in duration and cycles 2 to 12 are 21 days in duration.
  Using the Lugano Criteria for response assessment
Assessment of adverse events (eg. fatigue, diarrhoea, confusion, nausea, constipation, anaemia, dyspnoea) | Analysis of the adverse events will be completed in line with the primary and secondary endpoints; When all patients have completed 6 cycles of protocol treatment, when all patients have completed 12 cycles of treatment.
  Incidence, nature and severity of adverse events are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE).
Overall response rates (complete or partial response) to combination therapy. | At the end of combination therapy (cycle 12).Cycle 1 is 14 days in duration and cycles 2 to 12 are 21 days in duration.
  Using the Lugano criteria
Overall response rates | At the end of combination therapy (cycle 12). Cycle 1 is 14 days in duration and cycles 2 to 12 are 21 days in duration.
  Using the Lugano criteria
Absence of minimal residual disease (MRD) | Following six cycles and 12 cycles of combination treatment. Cycle 1 is 14 days in duration and cycles 2 to 12 are 21 days in duration.
  Measured by aggregate measure of peripheral blood and/or bone marrow flow cytometry, PCR and ctDNA
Progression-free survival (PFS) | Progression is measured from the date of registration to the date of first progression at any site or date of death due to any cause. Patients will be followed assessed until the last patient registered completes 5 years of follow up.
  Determined based on the modified Lugano criteria.
Duration of response | Patient's will be followed assessed until the last patient registered completes 5 years of follow up.
  Defined as the time from registration to date of death from any cause. Patients who have not died by the study close-out date will be censored at their last visit. Patients who are lost to follow-up before the close-out date and who are not known to have died will be censored at the date they were last known to be alive

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Centre, Parkville, Victoria
  - Sir Charles Gairdener, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared publicly. Aggregate patient data and final results will be presented in the final report.